CLINICAL TRIAL: NCT01641523
Title: Multicenter Prospective Controlled Study in Cranioplasty Reconstruction
Brief Title: Controlled Study in Cranioplasty Reconstruction
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Collaborators: Fin-Ceramica Faenza Spa (Industry)
Responsible Party: Principal Investigator, Franco Servadei, Franco Servadei, Prof. MD, Azienda Ospedaliero-Universitaria di Parma
Other Study IDs: NEU02
Record Dates: First submitted 2012-07-05; First posted 2012-07-16 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Cerebral Decompression Injury; Cranioplasty
Keywords: Cranioplasty prosthesis; Hydroxyapatite; PolyMethylMethacrylate; Autologous Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hydroxyapatite Cranioplasty: patient underwent to cranioplasty reconstruction with customized hydroxyapatite prosthesis
  Interventions: Device: CustomBone Service
- polymethylmethacrylate: patient underwent to cranioplasty reconstruction with polymethylmethacrylate prosthesis
  Interventions: Device: CustomBone Service
- autologous bone: patients underwent to cranioplasty reconstruction by autologous bone repositioning
  Interventions: Device: CustomBone Service

INTERVENTIONS:
Device: CustomBone Service — customized hydroxyapatite cranial prosthesis
  Other Names: polymethylmethacrylate cranioplasty; autologous bone opercula

SUMMARY:
Multicenter, prospective, comparative, observational study with regular follow-up visits.

The project's aim is long-term follow-up of patients affected by large and complex craniolacuniae treated, in standard clinical practice, with CustomBone Service™ Cranial (porous bio-mimetic hydroxyapatite custom-made medical device for cranioplasty), autologous bone or polymethilmethacrylate customized prosthesis and to compare the clinical outcome and safety among the three treatments.

Elegibility to each treatment will respect the standard clinical practice. Each investigator will respect his own hospital criteria for cranial reconstruction.

Each centre's agreement to participate the study is totally voluntary.

The study sample size has not been defined on statistical criteria: the study population was set at 100 consecutive patients treated with cranioplasty reconstruction with one of the three foreseen group.

Each investigator will not be allowed to enrol more then 20 patients to avoid an enrolment imbalance between centres involved.

Primary study end-points are: evaluation of adverse event incidence after surgical treatment.

Secondary end-points are: quality of life improvement, evaluation of bone continuity restoration evaluated by CT scan analysis, neurological improvement.

DETAILED DESCRIPTION:
Cranioplasty surgery is necessary everytime a craniolacuniae has to be reconstructed to ensure protection to the central nervous system. Cranioplasty surgery is classified into first line surgery, due to traumatic events or degenerative pathologies, and second line treatment, when due to first treatment failure, for example because of autologous bone reabsorption/infection or other material reject.

Clinical evaluation scores Specific and validated clinical scores will be employed for End-points evaluation.

CT scan will required in the pre-operation visit and in the post-operation time during the follow up visits to evaluate the bone-implant osteointegration process and osteointegration will be evaluated applying a specific score.

Data have been recorded in a e-CRF with limited access, protected by personal password.

Data will always be collected in an anonymous way, subjects identity will always be undisclosed.

Each patient will be asked to give informed consent to partecipate the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients which need cranial reconstruction,
2. Cranioplasty reconstruction by autologous bone, hidroxyapatite or polymethylmethacrylate,
3. Patients of both sex in age range between 14 and 75 years old,
4. Craniolacuniae size > 25 cm2 ,
5. Patients affected by complex pathologies or fracture or infection of a previous implant.
6. Elegibility to CustomBone Service™ Cranial treatment will respect the product leaflet instructions.
7. Each investigator will respect his own medical centre internal inclusion criteria to cranial reconstruction.

Exclusion Criteria:

1. Patients affected by important emocoagulation pathologies,
2. Patients affected by mellitus diabetes,
3. Patients affected by autoimmune pathology,
4. Patients unable to intend,
5. Patients affected by immunodepression.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: consecutive patients,in different italian centres, requiring cranioplasty
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2007-01; Primary Completion 2007-01 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Safety | 360 day after surgery
  incidence of adverse event (infection, reabsorption, mobilization, fractures, dislocation) after surgical treatment

SECONDARY OUTCOMES:
Efficacy | 90, 180, 360, 720 days after the surgery
  Quality of life improvement evaluation: Disability Rating Scale(DRS); Neurological recovery evaluation: Neurological Objective Exam (EON), Glasgow Coma Scale (GCS), Glasgow Outcome Scale (GCS), motor deficit evaluation scale; Mechanical, biological and aesthetic outcome; CT scan evaluation;

CONTACTS AND LOCATIONS:
Overall Officials: Franco Servadei, Prof. MD, Study Director — Maggiore Hospital Parma